CLINICAL TRIAL: NCT03202784
Title: A Phase 1, Single-Dose, 3-Period Crossover Study to Evaluate the Relative Bioavailability of Two BCX7353 Capsule Formulations and to Evaluate the Effect of Food on BCX7353 Pharmacokinetics in Healthy Subjects
Brief Title: A Relative Bioavailability Study of Two Formulations of BCX7353
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BCX7353-103
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2017-10

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Intervention Model Description: Three way crossover to evaluate two formulations of BCX7353 and to determine if there is a food effect
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCX7353 API in capsule (Experimental): fasted administration of BCX7353 API in capsule
  Interventions: Drug: BCX7353
- BCX7353 blend in capsule (Experimental): fasted administration of BCX7353 blend in capsule
  Interventions: Drug: BCX7353
- BCX7353 blend in capsule with food (Experimental): administration of BCX7353 blend in capsule following high-fat meal
  Interventions: Drug: BCX7353

INTERVENTIONS:
Drug: BCX7353 — BCX7353

SUMMARY:
This is an open-label, randomized study to investigate the relative bioavailability of two formulations of BCX7353 and to determine if there is a food effect

DETAILED DESCRIPTION:
In this study, 24 healthy subjects will be randomized to receive a single dose of two formulations of BCX7353 and one of the formulations administered with a high-fat meal. A 14-day washout period will separate each dose.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* acceptable birth control measures for male subjects and women of childbearing potential
* complies with all required study procedures and restrictions

Exclusion Criteria:

* clinically significant medical history, current medical or psychiatric condition
* clinically significant ECG finding, vital sign measurement or laboratory/urinalysis abnormality at screening or baseline
* current use, or use of any prescribed or over the counter medication, vitamins or herbal products within 14 days of Day 1
* participation in any other investigational drug study within 90 days of screening
* recent or current history of alcohol or drug abuse
* regular recent use of tobacco or nicotine products
* positive serology for HBV, HCV, or HIV
* pregnant or nursing
* donation or loss of greater than 400 mL of blood within the previous 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Geometric least-squares mean ratio for Cmax for test (blend in capsule) versus reference formulation (API in capsule) | plasma pharmacokinetic parameters are based on blood sampling over a 72 hour period
Geometric least-squares mean ratio for AUClast for test (blend in capsule) versus reference formulation (API in capsule) | plasma pharmacokinetic parameters are based on blood sampling over a 72 hour period
Geometric least-squares mean ratio for AUCinf for test (blend in capsule) versus reference formulation (API in capsule) | plasma pharmacokinetic parameters are based on blood sampling over a 72 hour period
Geometric least-squares mean ratio for Cmax for test (blend in capsule fed) versus reference formulation (blend in capsule fasted) | lasma pharmacokinetic parameters are based on blood sampling over a 72 hour period
Geometric least-squares mean ratio for AUClast for test (blend in capsule fed) versus reference formulation (blend in capsule fasted) | lasma pharmacokinetic parameters are based on blood sampling over a 72 hour period
Geometric least-squares mean ratio for AUCinf for test (blend in capsule fed) versus reference formulation (blend in capsule fasted) | lasma pharmacokinetic parameters are based on blood sampling over a 72 hour period

SECONDARY OUTCOMES:
adverse events | absolute and change from baseline through end of study, approximately 35 days
laboratory analyses | absolute and change from baseline through end of study, approximately 35 days
vital signs | absolute and change from baseline through end of study, approximately 35 days
physical examination findings | absolute and change from baseline through end of study, approximately 35 days
electrocardiograms | absolute and change from baseline through end of study, approximately 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB, BScMedSci, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom